CLINICAL TRIAL: NCT03974685
Title: Phase I Open Label Trial of Pharmacokinetics and Safety of 99mTc Niacinamide Polyethylene Glycol Bicyclic RGD Peptide (99mTc-3PRGD2) Injection in Healthy Volunteers
Brief Title: A Study of 99mTc-3PRGD2 Injection in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RDO Pharm. (Industry)
Collaborators: Beijing Pharbers Genesis Pharmaceutical Technology Co., Ltd. (Industry); MedAlly Solutions Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FSRDA201801
Record Dates: First submitted 2019-05-16; First posted 2019-06-05 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-05

CONDITIONS: Healthy
Keywords: 99mTc-3PRGD2; Integrin ανβ3; Dosimetry

STUDY DESIGN:
Intervention Model Description: Single Group Assignment drug:0.3mCi/kg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 99mTc-3PRGD2 (Experimental): Volunteers were injected intravenously and then scanned by SPECT/CT. Drugs use generic name：99mTc niacinamide polyethylene glycol bicyclic RGD peptide dosage form:Injection dosage:0.3mCi/kg frequency:single
  Interventions: Drug: 99mTc niacinamide polyethylene glycol bicyclic RGD peptide (99mTc-3PRGD2)

INTERVENTIONS:
Drug: 99mTc niacinamide polyethylene glycol bicyclic RGD peptide (99mTc-3PRGD2) — Single dose

SUMMARY:
The study drug 99mTc-3PRGD2 of this study is a new radioactive diagnostic preparation for clinical use as a nuclear medicine molecular probe for tumor SPECT/CT imaging.

After 99mTc-3PRGD2 is injected into the body, it is specifically taken up by integrin receptor-positive tumor tissue, and tumor tissue is developed by SPECT/CT, which can be used for molecular imaging diagnosis and individualized treatment of common tumors.

The primary objectives of this study is to examine the pharmacokinetics the safety of 99mTc-3PRGD2 injection in healthy volunteers, as well as the biodistribution in the human body and to estimate the dose of internal radiation absorbed. This study provides the basis for the design of phase II clinical research programs.

DETAILED DESCRIPTION:
To a large extent, cancer treatment outcomes depend on the accurate diagnosis and staging of the disease. An important basis for early diagnosis of malignant tumors is medical imaging. Single-Photon Emission Computed Tomography (SPECT) and Positron Emission Tomography (PET) are most well-developed nuclear medicine procedures based on the measurement of radiolabeled tracer molecules.

These radiotracers allow biologic processes to be measured and whole body images to be obtained, which will demonstrate exact locations of radiotracer accumulation. Functional imagings of SPECT and PET provide specific information which is not available from standard medical imaging modalities such as ultrasound, X-ray, computerized tomography (CT) or magnetic resonance imaging (MRI).

The test drug in this study is a new radioactive diagnostic preparation, consisting of radiochemical (Sodium Pertecheetate [99mTc] Injection) and a kit (including Three core ligands, HYNIC-3PRGD2, Tricine, TPPTS). Before administration, 99mTc:HYNIC-3PRGD2:Tricine:TPPTS (1:1:1:1) chelate compound (99mTc-3PRGD2) will be prepared as per standard opration presedure, which will be used as a molecular probe for SPECT/CT imaging.

The core ligand HYNIC-3PRGD2 is a novel RGD dimer that specifically binds to the integrin αvβ3 receptor with high selectivity and affinity. Integrin αvβ3 is highly expressed in tumor neovascularization. After injection, 99mTc-3PRGD2 will be specifically taken up by the integrin receptor-positive tumor tissue, then be imaged by SPECT/CT. The product can be used for molecular imaging diagnosis and individualized treatment for common tumors such as lung cancer and breast cancer are performed.

The primary objectives of this study is to examine the pharmacokinetics the safety of 99mTc-3PRGD2 injection in healthy volunteers, as well as the biodistribution in the human body and to estimate the dose of internal radiation absorbed. This study provides the basis for the design of phase II clinical research programs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers;
* 25 to 45 years of age, male to female ratio 1:1;
* Body mass index (BMI) ranges from 19 to 25 kg/m2 [Body mass index = body weight (kg)/ height squared (m2)];
* Clinical laboratory test results are normal, or laboratory values out of normal range is judged as not relevant for the clinical trial by the investigator;
* Subjects should read, sign an Informed Consent Form and willing to complete the trial according to the regulations.

Exclusion Criteria:

* Women who are breastfeeding or pregnant;
* Subjects with primary lesion in important organs;
* Subjects with mental or physical disorders;
* History of alcohol abuse or drug abuse;
* Subjects addict to coffee or smoker;
* Positive result on tests for HIV antibody, HbsAg or anti-hepatitis C virus antibody;
* History of allergic reactions to two or more kinds of drugs or foods or allergic to any components of test drug;
* Subjects with diseases (such as insomnia) are receiving other preventive/therapeutic drugs prior to study administration;
* Other reasons which, in the opinion of the investigator, would prevent the subject from participating in the study;
* Any anticipation in other clinical trial within 3 months;
* Subject received isotope treatment or examination before screening, or received X-ray examination more than three times within one year.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
AUC(0-t) | Day 1(dosing day )and Pre-dose,1,2,3,19,33,53,91,120,245 minutes post dose
  Area under the Activity-time curve from Hour 0 to the last measurable activity
The %ID(The radioactivity of the urine at each time period/ the total injection activity) | Day 1(dosing day)and Pre-dose,0-50 minutes,50-120 minutes,2-4 hours, 4-8 hours,8-12 hours,12-24hours post dose
  The %ID(The radioactivity of the urine at each time period/ the total injection activity) is calculated
The %ID(The radioactivity of the main organs at each time period/ the total injection activity) | post-intervention at 4 months
  The %ID(The radioactivity of the main organs at each time period/ the total injection activity) is calculated.
The radiation dosimetry of the test drug in organs | post-intervention at 4 months
  The internal radiation dosimetry (Dt,mSv) of each irradiated organ is calculated.
Radiochemical purity | During procedure
  To reflects the stability of the drug in the human body,that Radiochemical purity in urine and blood samples is measured.

SECONDARY OUTCOMES:
Incidence of adverse events | 3 days
  Assessment of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, professor, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No